CLINICAL TRIAL: NCT05367908
Title: Discoveries - Different Immunization Boosters for Covid-19: Effect on Response in Antibodies
Brief Title: A Study to Determine Antibody Levels After Receiving COVID-19 Boosters of Any Kind
Acronym: disCOVEries
Status: Completed | Type: Observational
Sponsor: ModernaTX, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: mRNA-1273-P914
Record Dates: First submitted 2022-05-06; First posted 2022-05-10 (Actual); Last update posted 2022-10-13 (Actual); Status verified 2022-10

CONDITIONS: SARS-CoV-2

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Cohort 1: MMM (Moderna Vaccine Series): Participants who have only received Moderna COVID-19 vaccines (that is, the 2-shot series and a booster).
- Cohort 2: PPP (Pfizer Vaccine Series): Participants who have only received Pfizer COVID-19 vaccines (that is, the 2-shot series and a booster).
- Cohort 3: V (Other Combination of Vaccines): Participants who have received any other combinations of boosters authorized in the United States, such as the 2-shot Pfizer series and a Moderna booster (PPM), the 2-shot Moderna series and a Pfizer booster (MMP), or the 1-shot Johnson and Johnson vaccine with either a Moderna or Pfizer booster.

SUMMARY:
This study will investigate antibody levels with respect to time since receiving a COVID-19 booster shot. The study will be decentralized, where participants can complete all study tasks at home. Self-reported participant information will be collected via surveys conducted at intake and monthly throughout the study. Participants will also perform monthly at-home capillary blood draws via YourBio devices that will be mailed to the designated laboratory for sample processing and antibody testing.

ELIGIBILITY:
Inclusion Criteria:

* Lives in the continental United States.
* Has been vaccinated against COVID-19 with a U.S.-authorized vaccine (that is, received the single shot J&J vaccine or both shots in the Pfizer or Moderna series).
* Has received a COVID-19 booster between September 2021 and screening.
* Is willing and able to submit vaccination card photo(s).
* Is willing and able to self-collect capillary blood 3 times during the study period via an at-home whole-blood collection device (that is, the YourBio TAP II Device).

Exclusion Criteria:

* Has been diagnosed with significant cognitive impairment or dementia.
* Has received more than one COVID-19 vaccine booster at screening.
* Is currently participating in a COVID-19 vaccine clinical trial.
* Is currently receiving chemotherapy or has received chemotherapy in the past 6 months.
* Is currently taking steroids, such as prednisone, for any condition.
* Has been diagnosed with or is taking medications for rheumatoid arthritis (RA), lupus or multiple sclerosis (MS).
* Has received an organ transplant
* Is currently undergoing dialysis of any kind (for example, hemodialysis or chronic ambulatory dialysis) for kidney disease.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Recruitment for this study will be aimed primarily at members of the Moderna Community on the Evidation platform. Evidation is an online platform where participants can connect digitally for educational health content, health data sharing, and research purposes. The study team will use an online strategy to invite, recruit, verify eligibility, consent, and enroll participants into this study. Potential participants will be provided a link to the study landing page on the Evidation platform, where they will be presented with an overview of the study. From the landing page, potential participants will be asked to complete a screening survey to determine participant eligibility and assess COVID-19 vaccination history to assist in cohort assignment.
Sampling Method: Non-Probability Sample
Enrollment: 1501 (Actual)
Dates: Start 2022-04-11 (Actual); Primary Completion 2022-08-14 (Actual); Study Completion 2022-08-14 (Actual)

PRIMARY OUTCOMES:
Change in Antibody Levels Since Receiving a COVID-19 Booster Vaccine at 0, 1, and 2 Months Post Enrollment | Baseline (Month 0), Month 1, and Month 2

CONTACTS AND LOCATIONS:
Locations (1):
- Evidation Health, San Mateo, California, United States